CLINICAL TRIAL: NCT03683823
Title: Efficacy of an Attention Guidance VR Intervention for Social Anxiety Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 the study was intitially paused and eventually ended.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-04-0011
Record Dates: First submitted 2018-07-20; First posted 2018-09-25 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-12

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention guidance (Experimental): In addition to the components included in the control intervention the experimental attention guidance condition consists of three unique components: (1) the rationale will include information about the importance of visually attending to the faces of the audience; (2) in addition to being given a speech topic, participants will be given target audience members to focus their gaze on during the speech. They will be told that they should look at and focus on the target audience member for the whole speech; (3) between speeches, the researcher will tell participants the percentage of time they were focused on the target face.
  Interventions: Behavioral: Attention guidance
- Control intervention (Active Comparator): Participants will complete two intervention sessions within one week. The intervention will use a manualized protocol.
  1. On the first session, participants will receive a brief standardized psychoeducation module, presented via a 15-minute video recording. This video will explain the intervention, its rationale, and the procedure.
  2. Participants will then have 5 minutes to plan and outline a speech based on a topic given to them. All participants will receive the same topic. Participants will not be allowed to use the outline during the public speaking exposure trials.
  3. Participants will then give six speeches that are each 3 minutes long on the same topic. Participants will give all the speeches in the immersive 360º-video environment.
  4. Between speeches participants will have a 1-minute break.
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Behavioral: Attention guidance — Explicitly guiding attention towards faces during public speaking exposures
  Arms: Attention guidance
Behavioral: Control intervention — Public speaking exposures
  Arms: Control intervention

SUMMARY:
Social anxiety disorder (SAD) is a prevalent mental health concern that impacts approximately 12% of the population. One mechanism thought to maintain SAD is avoidance of faces (i.e. avoidance of negative evaluative threat). However, research on attentional processes in SAD has been confined to paradigms presented on computer monitors. To investigate attentional processes in a more naturalistic way the investigators developed an immersive, 360º-video virtual reality environment using real actors, as part of a pilot study. Participants with a range of social anxiety symptoms (from none to severe) completed a 5-minute speech in this virtual reality environment while their eye movements were recorded. Results from the study showed that greater symptoms of social anxiety were associated with avoidance of looking at faces (i.e. fewer fixations on faces). While existing treatments for SAD are moderately effective, a large number of individuals do not experience meaningful reductions in their symptoms. The overarching goal of this project is inform future treatment research for SAD. The investigators will test a brief attention guidance intervention for SAD that specifically targets avoidance of faces as a potential mechanism maintaining the disorder. The proposed research will use the eye tracking hardware and naturalistic virtual reality environment from the pilot study. The investigators will also collect eye tracking data prior to the intervention in order to investigate potential heterogeneity in the attentional processes of SAD. The investigators will test the hypotheses that (a) the attention guidance intervention, compared to the control intervention, will result in a greater reduction in symptoms of social anxiety, and (b) this effect will be mediated by the number of fixations on faces during a brief public speaking challenge following the intervention. These results will provide causal evidence related to a hypothesized mechanism maintaining SAD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65;
2. Fluent in English;
3. Personal Report of Public Speaking Anxiety score > 98;
4. Leibowitz Social Anxiety Scale > 30;
5. Peak fear ≥ 50 on the behavioral approach task during the baseline assessment;
6. Meets DSM-5 Criteria for Social Anxiety Disorder.

Exclusion Criteria:

1. Currently receiving CBT for Social Anxiety Disorder;
2. Significant visual impairment precluding the use of virtual reality equipment;
3. Unstable dose of psychotropic medications within 3 weeks prior to baseline assessment;
4. Current alcohol or substance use disorders;
5. Current, or history of bipolar disorder; current, or history of psychosis;
6. Serious suicidal risk, as determined by clinical interview.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Intervention: Participants will complete two intervention sessions within one week. The intervention will use a manualized protocol.
  1. On the first session, participants will receive a brief standardized psychoeducation module, presented via a 15-minute video recording. This video will explain the intervention, its rationale, and the procedure.
  2. Participants will then have 5 minutes to plan and outline a speech based on a topic given to them. All participants will receive the same topic. Participants will not be allowed to use the outline during the public speaking exposure trials.
  3. Participants will then give six speeches that are each 3 minutes long on the same topic. Participants will give all the speeches in the immersive 360º-video environment.
  4. Between speeches participants will have a 1-minute break.
  Control intervention: Public speaking exposures
Period: Post-treatment Assessment
Arm/Group | Attention Guidance | Control Intervention
Started | 11 | 10
Completed | 10 | 8
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: 1-week Follow-up
Arm/Group | Attention Guidance | Control Intervention
Started | 10 | 8
Completed | 9 | 7
Not Completed | 1 | 1
Not completed — Research halted due to COVID-19 pandemic | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Guidance | Control Intervention | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.20 (1.23) | 25.90 (15.42) | 22.55 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
Personal Report of Public Speaking Anxiety [Mean (Standard Deviation); unit: score on a scale] — The range for the measure was 34-170, with higher values reflecting greater anxiety.
  score on a scale | 140.27 (16.85) | 139.40 (14.30) | 139.84 (15.58)
Liebowitz Social Anxiety Scale Self Report Version [Mean (Standard Deviation); unit: score on a scale] — The range for the measure was 0-144, with higher values reflecting greater anxiety.
  score on a scale | 75.27 (22.32) | 79.70 (25.64) | 77.49 (23.98)

OUTCOME MEASURES:

1. Primary Outcome: Personal Report of Public Speaking Anxiety Scale Post-intervention
Description: Questionnaire that assesses fear of public speaking Score range (total summed score): 34-170; Higher score reflects greater public speaking anxiety
Time Frame: Immediately following the end of the 1-week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Guidance | Control Intervention
Number analyzed (Participants) | 10 | 8
score on a scale | 123.50 (21.21) | 119.63 (19.54)

2. Primary Outcome: Personal Report of Public Speaking Anxiety Scale at 1-week
Description: Questionnaire that assesses fear of public speaking Score range: 34-170 (total summed score); Higher score reflects greater public speaking anxiety
Time Frame: 1-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Guidance | Control Intervention
Number analyzed (Participants) | 9 | 7
score on a scale | 123.56 (18.98) | 123.71 (17.01)

3. Secondary Outcome: Leibowitz Social Anxiety Scale Post-intervention
Description: Questionnaire that assesses generalized social anxiety Score range (total summed score): 0-144; Higher scores reflect greater social anxiety
Time Frame: Immediately following the end of the 1-week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Guidance | Control Intervention
Number analyzed (Participants) | 10 | 8
score on a scale | 64.80 (21.29) | 65.88 (27.27)

4. Secondary Outcome: Leibowitz Social Anxiety Scale at 1-week
Description: as for outcome 3
Time Frame: 1-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Guidance | Control Intervention
Number analyzed (Participants) | 9 | 7
score on a scale | 51.89 (28.18) | 55.57 (15.08)

5. Secondary Outcome: Speech Anxiety Thoughts Inventory Post-intervention
Description: Assesses cognitions associated with social anxiety Score range (total summed score): 23-115; Higher scores reflect greater severity
Time Frame: Immediately following the end of the 1-week intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Guidance | Control Intervention
Number analyzed (Participants) | 10 | 8
score on a scale | 73.80 (22.11) | 70.12 (19.69)

6. Secondary Outcome: Speech Anxiety Thoughts Inventory at 1-week
Description: as for outcome 5
Time Frame: 1-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Guidance | Control Intervention
Number analyzed (Participants) | 9 | 7
score on a scale | 64.22 (20.45) | 60.43 (18.30)

ADVERSE EVENTS:
Time Frame: Until study completion (approximately 2 weeks after the baseline assessment).
Description: The intervention was behavioral and well established to pose no risks.
Arm/Group | Attention Guidance | Control Intervention
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT03683823/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT03683823/SAP_001.pdf
  • Informed Consent Form (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT03683823/ICF_002.pdf